CLINICAL TRIAL: NCT01687283
Title: A Multicenter, Randomized, Single Blind, Active Controlled, Parallel Group Study to Determine Efficacy and Safety of Nebulized Fluticasone Propionate 1mg BID Compared With Nebulized Budesonide 2mg BID Administered for 12 Weeks in Chinese Adult and Adolescent Patients With Severe Persistent Asthma
Brief Title: Efficacy and Safety Study of Fluticasone Proponate Inhalation Solution in Adult and Adolescent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114219
Record Dates: First submitted 2012-08-23; First posted 2012-09-18 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Asthma
Keywords: fluticasone propionate inhalation solution; budesonide suspension for inhalation; efficacy; severe persistent asthma; pharmacokinetics; safety
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone propionate (Experimental): 1 mg BID inhalation via nebulizer
  Interventions: Drug: fluticasone propionate inhalation solution
- budesonide suspension (Active Comparator): 2 mg BID inhalation via nebulizer
  Interventions: Drug: budesonide suspension

INTERVENTIONS:
Drug: fluticasone propionate inhalation solution — 1 mg BID inhalation for 12 weeks with one possible chance to change to 0.5 mg BID
  Arms: fluticasone propionate
Drug: budesonide suspension — 2 mg BID inhalation for 12 weeks with one possible chance to change to 1 mg BID
  Arms: budesonide suspension

SUMMARY:
This is a multicentre, randomized, single-blind, active-controlled, parallel-group phase III local registration study for a treatment period of 12 weeks. This study aims to assess the effectiveness and safety of fluticasone propionate 1mg via nebulizer BID in treatment of Chinese adult and adolescent patients with severe persistent asthma for a treatment period of 12 weeks versus budesonide 2mg via nebulizer BID. The steady-state plasma pharmacokinetics of fluticasone propionate inhalation solution will also be assessed.

DETAILED DESCRIPTION:
Male or female subjects between 17 to 70 (inclusive) years of age with severe persistent asthma meeting the inclusion criteria and having completed the screening period of 2 weeks will, in a proportion of 1:1, randomly receive fluticasone propionate 1mg via nebulizer BID or budesonide 2mg via nebulizer BID for a treatment period of 12 weeks. The clinic visit will be arranged at 2 weeks, 4 weeks, 8 weeks and 12 weeks during study treatment. If the subjects meet the criteria of pre-defined asthma control at treatment 4 weeks or 8 weeks, they will have one chance to be treated with the half dose of study drug. 2 weeks after completion of study treatment or after early withdrawal from study, the follow-up visit will be performed to assess the post-treatment adverse events. The primary endpoint is the mean change from baseline in morning peak expiratory flow (PEF) over the 12 week treatment period. Safety assessments include adverse events, vital signs, oral and oropharyngeal candidiasis, hematological, biochemical tests), 24-hour urinary cortisol and 12-lead ECG. The steady-state plasma pharmacokinetics of fluticasone propionate inhalation solution will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female outpatients aged >=17 years and <=70 years
* A female is eligible to enter and participate in this study if she is:

Non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchal, post-menopausal), or Child-bearing potential, has a negative urinary pregnancy test at screening and agrees to take contraceptive precautions (including abstinence) (referring to appendix 1: Highly Effective Methods For Avoidance Of Pregnancy In Women Of Childbearing Potential) which, in the opinion of the investigator are adequate to prevent pregnancy during the study.

* A documented clinical history of asthma for a period of at least 12 weeks prior to Visit 1 based on the Guidance of Asthma Management and Prevention 2008 in China (refer to appendix 2).
* Demonstrated >=12% and >=200mL reversibility of FEV1 within 15-30minutes following inhalation of 200-400ug of salbutamol aerosol within 12 months prior to visit 1 or at the Screening Visit.
* Subjects have pre-bronchodilator FEV1% predicted between >=40% and <80% at visit 1.
* Subjects on a stable dose at least 2 weeks with high dose ICS (eg. Fluticasone Propionate 500ug twice daily or other ICS with equivalence doses, refer to Appendix 3) or moderate dose ICS plus LABA (eg. Fluticasone Propionate/Salmoterol 250/50ug , twice daily; or Budesonide/Formoterol Fumarate in maintainance160/4.5ug, two inhalation, twice daily; or other product equivalence doses).
* Subjects and/or their legally acceptable representative (if applicable) is willing to give informed consent to participate in the study, and having ability to comply with study procedures (including patients can use Nebulizer correctly, be able to understand and complete the diary cards and be able to record their PEF using a peak flow meter). The subjects and/or their legally acceptable representative (if applicable) will need to give additional informed consent to be eligible for blood pharmacokinetic samplings.

Exclusion Criteria:

* History of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of visit 1 and led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.
* Subjects have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the patient at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
* Subjects will not b eligible for the run-in if he/she has clinical visual evidence of candidias at visit 1.
* Current smoker or a smoking history of 10 pack years or more. A subject may not have used inhaled tobacco products (i.e., cigarettes, cigars or pipe tobacco) within the past 3 months.
* Patients who are pregnant or lactating.
* Patients having any known or suspected hypersensitivity to corticosteroids or the excipients of study drug, including Polysorbate 20, Sorbitan monolaurate, Monosodium phosphate dehydrate, Dibasic sodium phosphate anhydrous, Sodium Chloride and Water for Injection.
* Patients who have evidence of alcohol abuse.
* Patients who will have a pre-planned surgery operation in 6 months.
* Liver function tests: aspartate aminotransferase (AST) / alanine aminotransferase (ALT) >= 2 × upper limit of normal (ULN) or alkaline phosphatase (ALP) / bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Has QTc >= 450 msec or >= 480 msec for patients with bundle branch block at the time of screening.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating Investigator, sub Investigator, study coordinator, or employee of the participating Investigator.
* No subject is permitted to perform night shift work from Visit 1 until completion of the study treatment period.
* Use of the following medications within the following time intervals prior to visit 1 or during the study: Medication / No use within the following time intervals prior to Screening (Visit 1) or at any time during the study Systemic or oral corticosteroids / 2 weeks Depot corticosteroids /12 weeks Anti-IgE (e.g. Xolair)/ 12 weeks Oral long-acting beta2-agonists (e.g. bambuterol) and inhaled long-acting beta2-agonists (e.g. salmeterol, formoterol) or combination products containing inhaled long-acting beta2-agonists (e.g. Seretide, Symbicort) / 12 hours (the stable dose of ICS/LABA combination within 2 weeks prior to Visit 1 could be continued during the run-in period) Theophyllines, slow-release bronchodilators, anticholinergics, ketotifen, nedocromil sodium, sodium cromoglycate, Anti-leukotrienes including suppressors of leukotriene production and antagonists / 1 day Inhaled short-acting beta2-agonist / 4 hours (salbutamol will be supplied for rescue during the study) Potent Cytochrome P450 3A4 inhibitors(e.g. ritonavir, ketoconazole, itraconzole) / 4 weeks Prescription or over the counter medication that would significantly affect the course of asthma, or interact with sympathomimetic amines, such as: anticonvulsants (barbiturates, hydantoins, carbamazepine); polycyclic antidepressants; beta-adrenergic blocking agents; phenothiazines and monoamine oxidase (MAO) inhibitors /1 day Chinese traditional medicines used for treatment of asthma and other allergic diseases / 1 week Any other investigational drug / 30 days or within 5 half lives, whichever is longer

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2013-11-07 (Actual); Study Completion 2013-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- China (17):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Zhanjiang, Guangdong
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Xuzhou, Jiangsu
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Yinchuan, Ningxia
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Qingdao, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuxi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 317 Chinese adults and adolescents aged >= 17 years and <= 70 years with severe persistent asthma were planned to be enrolled in study. This study was conducted from 27-September-2012 to 7-November-2013.
Pre-assignment Details: Out of 460 screened participants, 109 were screen failures and 34 were run-in failures. Out of 317 participants, two participants did not receive the study drug and 315 participants received the study drug.
Groups:
- FP 1 mg BID: Participants received Fluticasone propionate (FP) oral inhalation (inhal) solution (sol'n) 1 milligram (mg) twice daily (BID) via nebulizer for a treatment period of 12 weeks. participants were allowed to use salbutamol aerosol inhaler for rescue of symptoms, and were followed-up for 2 weeks.
- BUD 2 mg BID: Participants received Budesonide (BUD) oral suspension for inhalation 2 mg BID via nebulizer for a treatment period of 12 weeks participants were allowed to use salbutamol aerosol inhaler for rescue of symptoms, and were followed-up for 2 weeks.
Period: Overall Study
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Started | 158 | 157
Completed | 123 | 130
Not Completed | 35 | 27
Not completed — Adverse Event | 11 | 4
Not completed — Lack of Efficacy | 3 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — protocol defined stopping criteria | 8 | 10
Not completed — Lost to Follow-up | 1 | 1
Not completed — Investigator discretion | 2 | 0
Not completed — Withdrawal by Subject | 9 | 8

BASELINE CHARACTERISTICS:
Population: The analysis was performed on intent-to-treat population. This population comprised of all participants randomized to treatment and who received at least one dose of study medication. Only the participants present at the indicated time point were analyzed.
Groups:
- FP 1 mg BID: Participants received FP oral inhalation solution 1 mg BID via nebulizer for a treatment period of 12 weeks. participants were allowed to use salbutamol aerosol inhaler for rescue of symptoms, and were followed-up for 2 weeks.
- BUD 2 mg BID: Participants received BUD oral suspension for inhalation 2 mg BID via nebulizer for a treatment period of 12 weeks participants were allowed to use salbutamol aerosol inhaler for rescue of symptoms, and were followed-up for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | FP 1 mg BID | BUD 2 mg BID | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (9.84) | 51.1 (6.65) | 51.4 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 71 | 148
  Male | 81 | 86 | 167
Region of Enrollment [Number; unit: Participants]
  China | 158 | 157 | 315

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 1 of Treatment Period/Visit 2) in Morning Peak Expiratory Flow (AM PEF) Over 12 Weeks in Intent-to-treat Population
Description: The peak expiratory flow (PEF) is a person's maximum speed of expiration, A peak flow meter was issued to participants at Visit 1 to measure the morning PEF prior to study drug and rescue medication. The best of three attempts was recorded by the participants in the diary cards. Baseline value was the assessment at Visit 2. The raw and change from baseline in daily AM PEF averaged over the 12-week treatment period The mean value was considered missing if less than 4 days were recorded in the baseline week prior to randomization or if less than 4 days are recorded after randomization. Analysis was performed using analysis of covariance (ANCOVA) model. Abbreviations used in statistical analysis section: standard deviation (SD) and significance (sig)
Time Frame: Baseline (Visit 2) and up to Week 12
Population: Intent-to-treat population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litres/Minute
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 155 | 152
Litres/Minute | 12.71 (3.677) | 14.51 (3.714)
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the lower limit of the two-sided 95% confidence interval for the treatment difference (FP minus BUD) in the mean change from baseline in daily AM PEF averaged over the 12 week treatment period was greater than -12 L/min; p = 0.733, ANCOVA — Analysis performed using ANCOVA with covariates of baseline, center, sex, age and treatment; Mean Difference (Net) = -1.80, 95% CI 2-sided [-12.19 to 8.59] — The analysis only included participants who had at least 4 days of non-missing AM PEF data in the baseline week prior to randomization and at least 4 days of non-missing AM PEF data after randomization

2. Primary Outcome: Change From Baseline (Day 1 of Trt Period/Visit 2) in AM PEF Over 12 Weeks in Per Protocol Population
Description: The peak expiratory flow (PEF) is a person's maximum speed of expiration, A peak flow meter was issued to participants at Visit 1 to measure the morning PEF prior to study drug and rescue medication. The best of three attempts was recorded by the participants in the diary cards. Baseline value was the assessment at Visit 2. The raw and change from baseline in daily AM PEF averaged over the 12-week treatment period The mean value was considered missing if less than 4 days were recorded in the baseline week prior to randomization or if less than 4 days are recorded after randomization. Analysis was performed using analysis of covariance (ANCOVA) model.
Time Frame: Baseline (Visit 2) and up to Week 12
Population: Per protocol population. This population comprised of all participants in the intent-to-treat Population who did not have any protocol violations which could impact treatment effect.Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litres/Minute
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 138 | 142
Litres/Minute | 13.50 (3.806) | 15.78 (3.750)
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.674, ANCOVA; Mean Difference (Net) = -2.28, 95% CI 2-sided [-12.95 to 8.38]

3. Secondary Outcome: Mean Change of Evening PEF From Baseline Over 12 Weeks
Description: The peak expiratory flow (PEF) is a person's maximum speed of expiration, A peak flow meter was issued to participants at Visit 1 to measure the evening PEF prior to study drug and rescue medication. The best of three attempts was recorded by the participants in the diary cards. Baseline value was the assessment at Visit 2. The raw and change from baseline in daily PM PEF averaged over the 12-weeks treatment period.
Time Frame: Baseline (Visit 2) and up to Week 12
Population: Intent-to-treat population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litres/Minute
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 156 | 153
Litres/Minute | 12.39 (3.469) | 15.16 (3.504)
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; Test type: Superiority or Other; p = 0.579, ANCOVA; Mean Difference (Net) = -2.77, 95% CI 2-sided [-12.57 to 7.04]

4. Secondary Outcome: Mean Change in Percentage of Symptom-free 24-hour Periods From Baseline Over 12 Weeks
Description: While calculating symptom-free 24-hour periods, a given 24-hour period was set to be "symptom free" only if the participant's responses to both the morning and evening assessments indicated no symptoms. The Baseline value was Visit 2 assessment and was derived from the last 7 days of the daily diary prior to the randomization. Change from Baseline was calculated as the difference between the value of the endpoint at the time point of interest and the baseline value. The value provided in outcome measure data is a consolidated value over Weeks 1 to 12.
Time Frame: Baseline (Visit 2) and over 12 Weeks
Population: Intent-to-treat population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hour
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 156 | 153
Percentage of symptom-free 24-hour | 21.77 (2.340) | 21.15 (2.364)
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; Test type: Superiority or Other; p = 0.854, ANCOVA; Mean Difference (Net) = 0.62, 95% CI 2-sided [-6.00 to 7.24]

5. Secondary Outcome: Median Day-time and Night-time Symptom Scores Per Participant Over 12 Weeks
Description: Participants recorded day-time symptom score every day in the morning and evening at bedtime before taking any rescue or study medication and before PEF measurement, using 6 point scale on Diary Card indicating 0 = No symptoms during the day and 5 =Symptoms so severe that participant could not go to work or perform normal daily activities. Night time symptoms were scored while waking in the morning on a scale of 0 (no symptoms) to 4 (severe). The value provided in outcome measure data is a consolidated value over Weeks 1 to 12.
Time Frame: Over 12 Weeks
Population: Intent-to-treat population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Score on Scale
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 156 | 153
Score on Scale
  Median day-time symptom score | 1.0 [0 to 4] | 1.0 [0 to 4]
  Median night-time symptom score | 1.0 [0 to 2] | 1.0 [0 to 3]
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; This statistical analysis is for comparison of FP 1 mg BID and BUD 2 mg BID in median day-time symptom score; Test type: Superiority or Other; p = 0.123, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: FP 1 mg BID vs BUD 2 mg BID; This statistical analysis is for comparison of FP 1 mg BID and BUD 2 mg BID in median night-time symptom score; Test type: Superiority or Other; p = 0.949, Wilcoxon rank sum test

6. Secondary Outcome: Mean Change in Percentage of Rescue-free 24-hour Periods From Baseline Over 12 Weeks
Description: While calculating rescue-free 24-hour periods, the 24-hour period was only set to be "rescue free" if responses to both the morning and evening, assessments indicated no use of rescue medication. If there were symptoms in either the morning or the evening then that 24-hour period was set to as "not symptom free". Similarly, if there was rescue medication use in either the morning or the evening, then that 24-hour period was set to as "not rescue free". The Baseline value was Visit 2 assessment and was derived from the last 7 days of the daily diary prior to the randomization. The value provided in outcome measure data is a consolidated value over Weeks 1 to 12.
Time Frame: Baseline and over 12 weeks
Population: Intent-to-treat population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue -free 24-hours
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 156 | 154
Percentage of rescue -free 24-hours | 19.27 (2.595) | 24.01 (2.612)
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; Test type: Superiority or Other; p = 0.204, ANCOVA; Mean Difference (Net) = -4.74, 95% CI 2-sided [-12.07 to 2.59]

7. Secondary Outcome: Median Number of Times Rescue Medication Use Over 12 Weeks
Description: Participants recorded the number of inhalations of rescue salbutamol inhalation aerosol used during the day and night. The baseline value was Visit 2 assessment and was derived from the last 7 days of the daily diary prior to the randomization. The analysis only included participants who had at least 2 days of non-missing numbers of times rescue medication (including zero) after randomization.
Time Frame: Up to week 12
Population: Intent-to-treat population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Number of Inhalations
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 156 | 153
Number of Inhalations | 0.0 [0 to 7] | 0.0 [0 to 4]
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; Test type: Superiority or Other; p = 0.170, Wilcoxon Rank sum

8. Secondary Outcome: Change of Clinical Lung Function Measurement Forced Expiratory Volume in One Second (FEV1) From Baseline Over 12 Weeks
Description: FEV1 as a measure of lung function assessment was measured at Week 2, 4, 8 and 12. FEV1 measures were performed electronically by spirometry. The highest of three technically acceptable measurements was recorded. FEV1 was measured prior to study drug administration and any rescue salbutamol use. Baseline value was the assessment at Visit 2.Change from baseline was calculated as the value at the specific time point minus baseline value.
Time Frame: Baseline and at Week 2, 4, 8 and 12
Population: Intent-to-treat population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | FP 1 mg BID | BUD 2 mg BID
Number analyzed (Participants) | 158 | 157
Litres
  Week 2: number analyzed (Participants) | 143 | 145
  Week 2 | 0.122 (0.0283) | 0.161 (0.0281)
  Week 4: number analyzed (Participants) | 128 | 134
  Week 4 | 0.187 (0.0333) | 0.195 (0.0328)
  Week 8: number analyzed (Participants) | 122 | 128
  Week 8 | 0.175 (0.0314) | 0.201 (0.0309)
  Week 12: number analyzed (Participants) | 117 | 126
  Week 12 | 0.217 (0.0342) | 0.200 (0.0336)
Statistical Analysis 1: Comparison: FP 1 mg BID vs BUD 2 mg BID; This statistical analysis is for comparison of FP 1 mg BID and BUD 2 mg BID in Change of clinical lung function measurement FEV1 at Week 2; Test type: Superiority or Other; p = 0.337, ANCOVA — Repeated Measures analysis adjusted for baseline, centre, sex, age, visit, treatment, visit by treatment interaction and visit by baseline interaction; Mean Difference (Net) = -0.039, 95% CI 2-sided [-0.118 to 0.041]
Statistical Analysis 2: Comparison: FP 1 mg BID vs BUD 2 mg BID; This statistical analysis is for comparison of FP 1 mg BID and BUD 2 mg BID in Change of clinical lung function measurement FEV1 at Week 4; Test type: Superiority or Other; p = 0.866, ANCOVA — Repeated Measures analysis adjusted for baseline, center, sex, age, visit, treatment, visit by treatment interaction and visit by baseline interaction; Mean Difference (Net) = -0.008, 95% CI 2-sided [-0.101 to 0.085]
Statistical Analysis 3: Comparison: FP 1 mg BID vs BUD 2 mg BID; This statistical analysis is for comparison of FP 1 mg BID and BUD 2 mg BID in Change of clinical lung function measurement FEV1 at Week 8; Test type: Superiority or Other; p = 0.566, ANCOVA — [p-value comment as in outcome 8, analysis 2]; Mean Difference (Net) = -0.025, 95% CI 2-sided [-0.113 to 0.062]
Statistical Analysis 4: Comparison: FP 1 mg BID vs BUD 2 mg BID; This statistical analysis is for comparison of FP 1 mg BID and BUD 2 mg BID in Change of clinical lung function measurement FEV1 at Week 12; Test type: Superiority or Other; p = 0.727, ANCOVA — [p-value comment as in outcome 8, analysis 2]; Mean Difference (Net) = 0.017, 95% CI 2-sided [-0.078 to 0.112]

9. Secondary Outcome: Steady-state Plasma Pharmacokinetics of Fluticasone Propionate Inhalation Solution- Time to Maximum Observed Plasma Concentration (Tmax)
Description: Tmax is defined as the time to maximum observed plasma concentration. Blood Pharmacokinetic (PK) samples were taken on Visit 3 (Day 14±2) pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose from participants. Blood sample for PK analysis, obtained within 72 hours of the last dose.
Time Frame: Pre-dose, 0.5 hour (h), 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose at Week 2
Population: Pharmacokinetics population included all participants whose PK samples were obtained and analyzed. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | FP 1 mg BID
Number analyzed (Participants) | 13
Hour | 0.905 (59.9)

10. Secondary Outcome: Steady-state Plasma Pharmacokinetics of Fluticasone Propionate Inhalation Solution-maximum Observed Plasma Concentration (Cmax)
Description: Cmax was defined as maximum observed plasma concentration. Blood PK samples were taken on Visit 3 (Day 14±2) pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose from participants. Blood sample for PK analysis, obtained within 72 hours of last dose.
Time Frame: Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose at Week 2
Population: Pharmacokinetic population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | FP 1 mg BID
Number analyzed (Participants) | 13
picogram per milliliter (pg/mL) | 59.24 (115.0)

11. Secondary Outcome: Steady-state Plasma Pharmacokinetics of Fluticasone Propionate Inhalation Solution-area Under the Plasma Concentration-time Curve for the Dose Interval [AUC (0-τ)]
Description: AUC (0-τ) was defined as the area under the plasma concentration-time curve for the dose interval. Blood PK samples were taken on Visit 3 (Day 14±2) pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose from participants. Blood sample for PK analysis, obtained within 72 hours of last dose.
Time Frame: Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose at Week 2
Population: Pharmacokinetic population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram hours per milliliter (pg*h/mL)
Arm/Group | FP 1 mg BID
Number analyzed (Participants) | 13
Picogram hours per milliliter (pg*h/mL) | 403.0958 (70.5)

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: Intent-to-treat population was used to assess adverse events up to Week 12.
Arm/Group | FP 1 mg BID | BUD 2 mg BID
All-Cause Mortality (participants affected / at risk) | 1/158 | 0/157
Serious Adverse Events (participants affected / at risk) | 4/158 | 2/157
Other Adverse Events (participants affected / at risk) | 23/158 | 15/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP 1 mg BID (N=158) | BUD 2 mg BID (N=157)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FP 1 mg BID (N=158) | BUD 2 mg BID (N=157)
Nasopharyngitis (Infections and infestations) | 13 | 10
Upper respiratory tract infection (Infections and infestations) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.